CLINICAL TRIAL: NCT06220227
Title: The Embryologist's Impact on Blastocyst Vitrification and Thawing: a Monocentric Retrospective Study With an External Validation Study.
Brief Title: The Embryologist's Impact on Blastocyst Vitrification and Thawing
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: EMBRYOFACTOR2
Record Dates: First submitted 2023-11-30; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Vitrification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- embryologist freezing the embryo
  Interventions: Procedure: vitrification and thawing procedures
- embryologist thawing the embryo
  Interventions: Procedure: vitrification and thawing procedures

INTERVENTIONS:
Procedure: vitrification and thawing procedures — Vitrification and thawing are crucial steps in infertility treatment. Vitrification solutions are aqueous cryoprotectant solutions that undergo solidification (and not freezing) when cooled at high rates to very low temperatures, thanks to an increase in viscosity.
  Thawing consists in remove the cryoprotectants, warm and dilute the blastocyst.

SUMMARY:
The goal of this monocentric retrospective observational study is to analyse, for the first time in literature, the role of the embryologist who freezes and thaws the embryos.

The primary objective of the study is to understand whether the embryologist who freezes and thaws the embryo influences the CPR (clinical pregnancy rate).

Secondary objectives, in case of statistically significant influence, are:

* Evaluate who influences more the CPR, between the embryologist who freezes the embryos and the embryologist who thaws the embryos.
* Evaluate if the embryologist who freezes and thaws the embryo impacts more than the embryologist or the physician who performs the ET.
* Evaluate whether the embryologists improve their performances, as their experience increases.
* Evaluate, through an external validation test, whether the model used can also be applied at other PMA centres

The study will consider all the freezing (vitrifications) and thawing procedures, performed at Humanitas Fertility Center between January 2019 and June 2023.

The study will include the transfers of single blastocysts, cryopreserved at Humanitas Fertility Center. On the other hand, the blastocysts transferred from other centres and the donor blastocysts will be excluded from the study, as well as multiple blastocysts transfers and the LP cycles.

The embryologist's experience will be assessed in terms of number of previous cryopreservation (vitrification) and thawing procedures. We will include in the study all the embryologists who performed at least 50 freezing and thawing.

For the evaluation of the study objectives, data will be gathered using a specific internal web-based database.

The final model will be created by analysing the Humanitas Fertility Center dataset and validated using datasets extrapolated from similar population from the San Raffaele Hospital infertility centre

ELIGIBILITY:
Inclusion Criteria:

The study database will include all the patients who performed a single cryopreserved blastocyst transfer, between January 2019 and June 2023, including also PGTA and repeated ART cycles.

The embryologist's experience will be assessed in terms of number of previous cryopreservation (vitrification) and thawing procedures. We will include in the study all the embryologists who performed at least 50 freezing and thawing.

Exclusion Criteria:

The blastocysts transferred from other centres and the donor blastocysts will be excluded from the study, as well as multiple blastocysts transfers and the LP cycles, to reduce the risk of selection bias or physician-embryologist couple bias.

The embryologists who performed less than 50 freezing and thawing will be excluded from the study.

Similarly, the first 50 procedures performed by each embryologist will not be counted in the data set.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study sample will include all the embryologists who freeze and thawed the embryos used for ART cycles at Humanitas Fertility Center between January 2019 and June 2023, matching the inclusion and exclusion criteria cited above.
Sampling Method: Probability Sample
Enrollment: 6800 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
clinical pregancy rate | January 2019-June 2023
  visualisation of the gestation sac in the uterus by ultrasound over the number of ET cycles performed

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy